CLINICAL TRIAL: NCT01061346
Title: Effect of Dietary Fat When Eaten With Fructose vs. Glucose on Insulin Resistance and Liver Fat
Brief Title: Effect of Dietary Fat When Eaten With Fructose Versus Glucose
Acronym: Fructose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, George A. Bray, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 29025
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Body Weight Changes
Keywords: Fructose; Glucose
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Fat Diet with Fructose (Experimental): 40% fat, 45% carbohydrate (with 20% fructose beverage), 15% protein
  Interventions: Other: 40% Fat Diet, 20% Fructose Beverage
- High Fat Diet with Glucose (Experimental): 40% fat, 45% carbohydrate (with 20% glucose beverage), 15% protein
  Interventions: Other: 20% Glucose Beverage
- Low Fat Diet with Glucose (Experimental): 20% fat, 65% carbohydrate (with 20% glucose beverage), 15% protein.
  Interventions: Other: 20% Glucose Beverage

INTERVENTIONS:
Other: 40% Fat Diet, 20% Fructose Beverage — 40% fat, 45% carbohydrate (with 20% fructose beverage), 15% protein
  Other Names: Fructose vs. Glucose
  Arms: High Fat Diet with Fructose
Other: 20% Glucose Beverage — 40% fat, 45% carbohydrate (with 20% glucose beverage), 15% protein
  Other Names: Fructose vs. Glucose
  Arms: High Fat Diet with Glucose
Other: 20% Glucose Beverage — 20% fat, 65% carbohydrate (with 20% glucose beverage), 15% protein
  Other Names: Fructose vs Glucose
  Arms: Low Fat Diet with Glucose

SUMMARY:
This study is designed to test the effects on liver fat of varying fat intake in the presence of fructose or glucose. We hypothesize that higher dietary fat when eaten with fructose as compared to glucose will increase the amount of hepatic lipid as measured by magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
After 2 screening visits including an exercise test, DEXA and CT scan, qualifiers begin a 7 day diet with 20% fat, 65% carbohydrate (with 20% glucose) and 15 % protein. Participants consume 2 meals per day at PBRC with lunch and weekend meals packed to go. Following a test day, participants are randomized to one of 3 diet assignments and then test again:

1)20% fat, 65% carbohydrate (with 20% glucose beverage), 15% protein 2)40% fat, 45% carbohydrate (with 20% glucose beverage), 15% protein 3)40% fat, 45% carbohydrate (with 20% fructose beverage), 15% protein On Day 7 and again 14 days later participants have labs, an oral Glucose tolerance test, hepatic and intramuscular lipid measures by MRS, vital signs and waist measurement.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 kg/m2 inclusive
* At least one of the following:

  1. Impaired fasting glucose between 100-125 mg/dl inclusive
  2. HDL below 40 mg/dl for men or below 50 mg/dl for females
  3. Triglycerides between 150 mg/dl and 400 mg/dl inclusive
  4. Blood pressure above or equal to 135 / 85 mm Hg
* Waist circumference >94cm (37 inches) for men or >80cm for women
* Mainly Healthy

Exclusion Criteria:

* Unable or unlikely to eat study foods and only foods provided by PRBC
* Taking routine medications except birth control pills
* Smoke, Abuse drugs,or Alcohol
* Pregnant or breastfeeding, irregular menstrual cycles, Post-menopausal,or PCOS
* Diabetes, heart, lung, liver, blood, or Kidney disease

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evidence to determine whether intake in beverages that provide 20% fructose or a similar beverage made with glucose given with a higher fat diet has an effect on your body weight, blood pressure, fats in your liver or your blood sugar. | One Month

CONTACTS AND LOCATIONS:
Overall Officials: George A Bray, MD, Principal Investigator — Pennington Biomedical Research Center; Sudip Bajpcyi, PhD, Study Chair — Pennington Biomedical Research Center
Locations (1):
- Pennintgon Biomedical Research Center, Baton Rouge, Louisiana, United States